CLINICAL TRIAL: NCT00262054
Title: Prospective, Randomized, Double-Blind, Active-Controlled, Multicenter Trial of Bivalirudin and Un-fractionated Heparin in Patients Undergoing Percutaneous Coronary Interventions. ISAR-REACT-3
Brief Title: Un-fractionated Heparin Versus Bivalirudin During Percutaneous Coronary Interventions (PCI) (ISAR-REACT-3)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Prof. A. Schömig, Deutsches Herzzentrum Munich
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GE IDE No. A01005; KKF 1.1-05
Record Dates: First submitted 2005-12-05; First posted 2005-12-06 (Estimated); Last update posted 2010-03-15 (Estimated); Status verified 2008-08

CONDITIONS: Coronary Disease; Angina Pectoris
Keywords: coronary disease
MeSH Terms: conditions — Coronary Disease; Angina Pectoris | interventions — bivalirudin; Abciximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): bivalirudin is to be administered as an intravenous bolus of 0.75 mg/kg prior to the start of the intervention, followed by infusion of 1.75 mg/kg per hour for the duration of the procedure.
  Interventions: Drug: Bivalirudin
- B (Active Comparator): UFH given as an intravenous bolus of 140 units/kg. Double blinding will be maintained by using a double-dummy technique consisting of identical UFH and bivalirudin syringes and bivalirudin or placebo infusion bags.
  Interventions: Drug: Un-fractionated heparin

INTERVENTIONS:
Drug: Bivalirudin — bivalirudin to be administered as an intravenous bolus of 0.75 mg/kg prior to the start of the intervention, followed by infusion of 1.75 mg/kg per hour for the duration of the procedure.
  Other Names: ReoPro
  Arms: A
Drug: Un-fractionated heparin — UFH is given as an intravenous bolus of 140 units/kg followed by infusion of placebo 1.75 mg/kg per hour for the duration of the procedure.
  Arms: B

SUMMARY:
The purpose of this study is to determine whether bivalirudin given during PCI is associated with better outcomes compared to un-fractionated heparin.

DETAILED DESCRIPTION:
Thrombin plays a major role in acute coronary artery occlusions during percutaneous coronary interventions. Unfractionated heparin has been traditionally used during invasive coronary procedures to reduce the risk of thrombotic occlusion. Bivalirudin, a direct antithrombin inhibitor, has several advantages over unfractionated heparin: it acts independently of antithrombin and inhibits both free and clot-bound thrombin; it is not neutralized by circulating inhibitors; exhibits consistent dose-response characteristics, and does not cause thrombocytopenia. Previous studies have shown that use of bivalirudin among patients undergoing percutaneous coronary interventions is associated with better outcomes (death, myocardial infarction, urgent repeat revascularization or in-hospital major bleeding) as compared with unfractionated heparin and adjunctive use of glycoprotein IIb/IIIa platelet receptor inhibitors. However, previous studies have included patients treated with plain balloon angioplasty or stenting after inadequate pre-treatment with thienopyridines (ticlopidine or clopidogrel). Recent guidelines recommend that all patients undergoing percutaneous coronary interventions must receive a loading dose of 300 -600 mg of clopidogrel. A 600 mg loading dose of clopidogrel eliminates the need for glycoprotein IIb/IIIa platelet receptor inhibitors in adjunct to heparin. According to existing evidence antithrombotic regimens based on either bivalirudin or pre-treatment with 600 mg of clopidogrel in addition to UFH intraprocedurally, are effective strategies to reduce ischemic and hemorrhagic complications in patients with coronary artery disease undergoing PCI. At present, it is not known whether bivalirudin is superior to UHF in patients who have been optimally pre-treated with a loading dose of clopidogrel.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age to undergo PCI
* Clopidogrel loading at least 2 hrs prior to PCI according to the PCI guidelines
* Informed, written consent

Exclusion Criteria:

* Recent ST-elevation myocardial infarction within the last 48 hours
* Cardiogenic shock
* ACS and positive biomarkers (Troponin T > 0.03 µg/L)
* Malignancies or other comorbid conditions (for example severe liver, renal and pancreatic disease) with life expectancy less than one year or that may result in protocol non-compliance
* Active bleeding; bleeding diathesis
* History of gastrointestinal or genitourinary bleeding within the last 6 weeks
* Presence of diseases which have a high probability of vascular lesions and subsequent bleeding such as active gastric ulcer or active ulcerous colitis
* Recent trauma or major surgery in the last month
* Ophthalmic surgery or brain surgery in the last month
* Retinopathies or vitreous body bleeding in the last month
* History of intracranial bleeding or structural abnormalities (for example aneurysm of cerebral arteries)
* Suspected aortic dissection; pericarditis and subacute bacterial endocarditis
* Patient's refusal to blood transfusion
* Oral anticoagulation therapy with coumarin derivative within the last 7 days
* Treatment with UFH within 6 hours or low-molecular weight heparin within 8 hours before randomization
* Treatment with bivalirudin within 24 hours before randomization
* Severe uncontrolled hypertension >180/110 mmHg unresponsive to therapy
* Planned staged PCI procedure within 30 days from index procedure or prior PCI within the last 30 days
* Relevant hematologic deviations:hemoglobin < 100 g/L; platelet count < 100 x 109 /L
* Glomerular filtration rate (GFR) < 30 ml/min or serum creatinine > 30 mg/L or dependence on renal dialysis
* Known allergy to the study medications: aspirin, clopidogrel, UFH, bivalirudin; stainless steel; true anaphylaxis after prior exposure to contrast media
* Known heparin-induced thrombocytopenia (Typ II)
* Previous enrollment in this trial
* Pregnancy (present, suspected or planned) or positive pregnancy test
* Spinal, peridural and epidural anesthesia
* Patient's inability to fully cooperate with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4570 (Actual)
Dates: Start 2005-11; Primary Completion 2008-02 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Composite rate of death, myocardial infarction (MI),urgent target vessel revascularization (TVR) within 30 days or in-hospital major bleeding | 30 days

SECONDARY OUTCOMES:
Composite rate of death, MI or urgent TVR within 30 days | 30 days
Composite rate of death, MI or TVR at 1 year | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Albert Schomig, MD, Study Chair — Deutsches Herzzentrum Muenchen; Adnan Kastrati, MD, Principal Investigator — Deutsches Herzzentrum Muenchen; Franz-Josef Neumann, MD, Study Director — Herz-Zentrum Bad Krozingen
Locations (4):
- Germany (4):
  - Herz-Zentrum, Bad Krozingen
  - Segeberger Kliniken, Bad Segeberg
  - Deutsches Herzzentrum Muenchen, Munich
  - First Medizinische Klinik, Klinikum rechts der Isar, Munich

REFERENCES:
- [Background] Verstraete M. Direct thrombin inhibitors: appraisal of the antithrombotic/hemorrhagic balance. Thromb Haemost. 1997 Jul;78(1):357-63. No abstract available. PMID 9198179
- [Background] Lincoff AM, Bittl JA, Harrington RA, Feit F, Kleiman NS, Jackman JD, Sarembock IJ, Cohen DJ, Spriggs D, Ebrahimi R, Keren G, Carr J, Cohen EA, Betriu A, Desmet W, Kereiakes DJ, Rutsch W, Wilcox RG, de Feyter PJ, Vahanian A, Topol EJ; REPLACE-2 Investigators. Bivalirudin and provisional glycoprotein IIb/IIIa blockade compared with heparin and planned glycoprotein IIb/IIIa blockade during percutaneous coronary intervention: REPLACE-2 randomized trial. JAMA. 2003 Feb 19;289(7):853-63. doi: 10.1001/jama.289.7.853. PMID 12588269
- [Background] Silber S, Albertsson P, Aviles FF, Camici PG, Colombo A, Hamm C, Jorgensen E, Marco J, Nordrehaug JE, Ruzyllo W, Urban P, Stone GW, Wijns W; Task Force for Percutaneous Coronary Interventions of the European Society of Cardiology. Guidelines for percutaneous coronary interventions. The Task Force for Percutaneous Coronary Interventions of the European Society of Cardiology. Eur Heart J. 2005 Apr;26(8):804-47. doi: 10.1093/eurheartj/ehi138. Epub 2005 Mar 15. PMID 15769784
- [Background] Kastrati A, Mehilli J, Schuhlen H, Dirschinger J, Dotzer F, ten Berg JM, Neumann FJ, Bollwein H, Volmer C, Gawaz M, Berger PB, Schomig A; Intracoronary Stenting and Antithrombotic Regimen-Rapid Early Action for Coronary Treatment Study Investigators. A clinical trial of abciximab in elective percutaneous coronary intervention after pretreatment with clopidogrel. N Engl J Med. 2004 Jan 15;350(3):232-8. doi: 10.1056/NEJMoa031859. PMID 14724302
- [Result] Schulz S, Mehilli J, Ndrepepa G, Neumann FJ, Birkmeier KA, Kufner S, Richardt G, Berger PB, Schomig A, Kastrati A; Intracoronary Stenting and Antithrombotic Regimen: Rapid Early Action for Coronary Treatment (ISAR-REACT) 3 Trial Investigators. Bivalirudin vs. unfractionated heparin during percutaneous coronary interventions in patients with stable and unstable angina pectoris: 1-year results of the ISAR-REACT 3 trial. Eur Heart J. 2010 Mar;31(5):582-7. doi: 10.1093/eurheartj/ehq008. Epub 2010 Feb 11. PMID 20150324
- [Result] Kastrati A, Neumann FJ, Mehilli J, Byrne RA, Iijima R, Buttner HJ, Khattab AA, Schulz S, Blankenship JC, Pache J, Minners J, Seyfarth M, Graf I, Skelding KA, Dirschinger J, Richardt G, Berger PB, Schomig A; ISAR-REACT 3 Trial Investigators. Bivalirudin versus unfractionated heparin during percutaneous coronary intervention. N Engl J Med. 2008 Aug 14;359(7):688-96. doi: 10.1056/NEJMoa0802944. PMID 18703471